CLINICAL TRIAL: NCT04891068
Title: BRE-04: Window of Opportunity Trial of Preoperative Low Dose Azacitidine in High-Risk Early Stage Breast Cancer
Acronym: BRE-04
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Vijayakrishna Krishnamurthy Gadi, Prinicpal Investigator, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0215
Record Dates: First submitted 2021-05-11; First posted 2021-05-18 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer Invasive; Early-stage Breast Cancer; High Risk Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — Azacitidine

STUDY DESIGN:
Intervention Model Description: Single arm, window of opportunity trial in which patient with previously untreated high risk early stage breast cancer will receive 5 consecutive days of azacitidine 50mg/m2 SC followed by standard of care therapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm with previously untreated high risk early stage breast cancer (Experimental): All participants will receive azacitidine 50mg/m2 SC daily for five consecutive days.
  Interventions: Drug: Azacitidine

INTERVENTIONS:
Drug: Azacitidine — 5-Azacitidine is a pyrimidine nucleoside analog in which nitrogen replaces carbon at position 5
  Other Names: Vidaza

SUMMARY:
To determine the effect of low dose azacitidine therapy on tumor infiltrating lymphocytes (TILs) in primary tumors from patients with high-risk early stage breast cancer, paired t-tests will be first used to compare TIL count in pre- and post-treatment specimens.

DETAILED DESCRIPTION:
To determine the effect of low dose azacitidine therapy on tumor infiltrating lymphocytes (TILs) in primary tumors from patients with high-risk early stage breast cancer, paired t-tests will be first used to compare TIL count in pre- and post-treatment specimens. Median TIL counts will be compared between the pre- and post-treatment specimens with the Wilcoxon signed-rank test if TIL count does not follow normal distribution. General linear model (GLM) or kruskal wallis test will be used in the multivariate analyses to estimate the effect of low dose azacitidine therapy on TILs after adjusting for other clinical factors and patients characteristics, including the heterogeneity of tumors.

Screening Evaluation Visit All screening procedures will take place within 30 days of the first treatment visit unless otherwise noted.

* Informed consent, HIPAA authorization
* Medical history including prior and concurrent therapies and pathology
* Physical exam, height, weight
* Vital signs (blood pressure, heart rate, temperature)
* Review of concomitant medications
* ECOG performance status
* Blood chemistries (sodium, potassium, serum creatinine [or GFR], calcium, albumin, ALT, AST, total bilirubin, alkaline phosphatase, total protein)
* CBC with differential
* Hepatitis B screening (hepatitis B surface antigen (HBsAg), hepatitis B core antibody (anti-HBc), total Ig or IgG, and antibody to hepatitis B surface antigen (anti-HBs))
* Diagnostic Mammogram (NOTE: can be performed up to 60 days prior to study enrollment) Tumor and axillary assessment
* Surgical assessment
* Serum pregnancy test for women of childbearing potential (NOTE: serum βhCG within 14 days prior to study registration).
* Archival tumor tissue assessment

Azacitidine Treatment Visits Day 1

* Pre-treated with ondansetron 8mg PO once 30 minutes prior to azacitidine administration.
* Urine pregnancy test for women of childbearing-potential (NOTE: if >7days since screening)
* Research blood draw
* Azacitidine administration
* AE assessment

Days 2-5

* Premedicate with ondansetron 8mg PO once 30 minutes prior to azacitidine administration.

  * Azacitidine administration

Pre study biopsy visit

* Physical exam, weight
* Vital signs (blood pressure, heart rate, temperature)
* Review of concomitant medications
* ECOG performance status
* Blood chemistries (sodium, potassium, serum creatinine [or GFR], calcium, albumin, ALT, AST, total bilirubin, alkaline phosphatase, total protein)
* CBC with differential
* Research blood draw
* AE assessment

Post Study Biopsy Follow-Up visit

* Physical exam, weight
* Vital signs (blood pressure, heart rate, temperature)
* Review of concomitant medications
* ECOG performance status
* Research blood draw
* Archival tumor tissue assessment
* AE assessment

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years of age at time of consent
2. ECOG 0, 1, or 2
3. Histologically confirmed invasive breast carcinoma documented by biopsy. AJCC 8th edition clinical stage T1a-T3/N0-N1/M0 by physical exam or radiologic studies
4. Disease characteristics I. TNBC (Less than or equal to 10% of tumor cells staining for ER and for PR by immunohistochemistry (IHC). HER2-negative, as defined by ASCO/CAP guidelines)

OR

II. ER positive (as determined by immunohistochemistry (IHC)) and any of the following high risk characteristics:

1. HER2 positive (IHC or FISH)
2. Node positive
3. Any clinical high-risk expression profile (mammaprint, oncotype, endopredict)
4. PR negative (IHC) OR III. HER 2 positive (as defined by ASCO/ACP guidelines) f. Demonstrates adequate organ function as defined in table below. All screening labs to be obtained within 30 days prior to registration.

System Laboratory Value Hematological Leukocytes ≥3,000/mm3 Platelet count ≥ 100,000/mm3 Absolute Neutrophil Count (ANC) ≥ 1,500/mm3 Hemoglobin (Hgb) ≥ 9.0 g/dL Renal Creatinine/Calculated creatinine clearance (CrCl) Cr < 1.5 x upper limit of normal (ULN) or CrCl ≥ 50 mL/min using the Cockcroft-Gault formula Hepatic Bilirubin Bilirubin ≤ 1.5 × ULN. Subjects with Gilbert's syndrome may have a bilirubin > 1.5 × ULN, if no evidence of biliary obstruction exists Aspartate aminotransferase (AST) ≤ 2.5 × ULN Alanine aminotransferase (ALT) ≤ 2.5 × ULN g. No evidence of distant metastases (M0 per AJCC staging guidelines) h. Provided written informed consent and HIPAA authorization for release of personal health information, via an approved UIC Institutional Review Board (IRB) informed consent form and HIPAA authorization.

i. Women of childbearing potential must not be pregnant or breast-feeding. A negative serum or urine pregnancy test is required per institutional practice guidelines.

j. As determined at the discretion of the enrolling physician or protocol designee, ability of the subject to understand and comply with study procedures for the entire length of the study.

Exclusion Criteria:

1. Previous anti-cancer treatment (cytotoxic chemotherapy, immunotherapy, biologic therapy, radiotherapy directed towards the primary breast tumor and/or ipsilateral axillary lymph nodes or investigational agents) with therapeutic intent for the current breast cancer.
2. Any type of breast implants
3. Active infection requiring systemic therapy
4. Uncontrolled HIV/AIDS or active viral hepatitis
5. Pregnant or nursing
6. Any prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of this investigational regimen, as determined by the treating medical oncologist.
7. Any mental or medical condition that prevents the patient from giving informed consent or participating in the trial unless a Legal Authorized Representative (LAR) is in place to sign on behalf of the patient.
8. Other major comorbidity, as determined by study PI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-01-10 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change in tumor infiltrating lymphocytes (TILs) count in primary tumors from patients with high-risk early stage breast cancer following low-dose azacitidine therapy. | 2 weeks from first dose of azacitidine
  Number of participants that show tumor infiltrating lymphocytes (TILs) in primary tumors from patients with high-risk early stage breast cancer

SECONDARY OUTCOMES:
Clinical response (change Ki67 and tumor size) of primary tumor following treatment with low dose azacitidine therapy | 2 weeks from first dose of azacitidine
  Number of participants that have a clinical response at time of surgery based on changes in the Ki-67 index
Safety - completion rate of low-dose azacitidine | 30 days after last dose of azacitidine
  Number of participants that fail to complete the planned course of treatment intervention using the NCI Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 5
Safety - tolerability of low-dose azacitidine therapy assessed by using the NCI Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 5 | 30 days after last dose of azacitidine
  Number of participants that have treatment related adverse events using the NCI Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 5
Disease Free Survival (DFS) | 2 years
  Number of days participants had DFS
Overall Survival (OS) | 2 years
  Number of days participants had OS

CONTACTS AND LOCATIONS:
Overall Officials: Vijayakrishna Krishnamurthy Gadi, MD, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois Cancer Center, Chicago, Illinois, United States